CLINICAL TRIAL: NCT06954272
Title: Characterisation of Skin Microstructure Under Normal and Atrophied States
Acronym: COSMOS
Status: Recruiting | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH23036
Record Dates: First submitted 2024-05-03; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Participants with healthy skin and no history of skin diseases with the exception of acne.
- Atopic dermatitis: Participants with atopic dermatitis and signs of adverse skin changes caused by topical corticosteroid use.

SUMMARY:
Skin dermatoses are a major health concern around the world, with heavy economic, social, and psychological burdens. Due to their chronic and incurable nature, they are serious diseases that cause physical pain in patients and reduced quality of life. Atopic dermatitis is the most common inflammatory skin disease with a prevalence of almost 20% in children and 10% in adults. Current therapies are designed to control the condition rather than cure it. Therefore, these therapies are lifelong and, when the disease is flaring, must be used intensively to achieve control. Despite the emergence of various therapies, topical corticosteroids (TCS) remains the gold standard therapy generally used as a first-line treatment. However, if used inappropriately, it can act like a double-edged sword. With the beneficial action of TCS comes the potential for undesirable effects, like skin thinning, especially when used long-term or excessively.

The objective of this study is to define the normal structural parameters for healthy skin in a diverse cohort, determine the effect of age, sex, and ethnicity and subsequently study how these values differ in clinically abnormal skin resulting from excessive or inappropriate use of topical corticosteroids (TCS). This will be achieved by using optical coherence tomography (OCT) to non-invasively image the skin. By undertaking this study, the investigators will gain real-world insight into the effects of long-term TCS use on the skin.

DETAILED DESCRIPTION:
Around 24% of the United Kingdom (UK) population seeks medical attention regarding a skin condition each year, of which 6.1% are referred to specialist dermatology care. Skin conditions are the most common reason for people to consult their General Practitioner (GP) (average of 630 consultations per GP every year). The most common skin conditions include eczema, psoriasis, acne, rosacea and urticaria. All are chronic inflammatory conditions with complex aetiology that require regular treatment (there is no cure). Each of these conditions has a significant impact on quality of life, with that impact being similar to epilepsy, asthma, cystic fibrosis, and renal disease for eczema, urticaria and psoriasis. Beyond new treatments, new ways of characterising these conditions are needed to better inform treatment decisions (treatment choice and regimen) and improve long-term management.

Recent research has demonstrated the potential of OCT to visually characterise skin inflammation. Conceptually similar to ultrasound, OCT uses light instead of sound to generate volumetric scans of the skin. With an axial resolution of <5 µm and a penetration depth of <2mm, cross-sectional images of the skin are comparable to tissue sections obtained via biopsy. In addition to enabling the quantification of the structural features of the skin, further processing can be used to derive detailed angiographs of the superficial dermal vasculature and birefringence patterns associated with dermal collagen structure. Several interesting metrics can be derived from OCT images, including epidermal thickness, depth of the superficial plexus, diameter of blood vessels, density of the vascular network, and index of collagen matrix. Through the investigating team's work on the Skin Pathology assessment with Optical Technologies (SPOT) study, a strong association between OCT-derived metrics like this and disease severity at specific anatomical locations (the cubital fossae) has been revealed in Atopic dermatitis (AD) patients. These metrics can be used to objectively assess the severity of eczema. In addition to enabling rapid and non-invasive monitoring of treatment efficacy (normalisation of skin structure) over time, they can also be used to quantify the adverse effects of inappropriate or excessive treatment. For example, the investigators have previously shown that continued use of topical corticosteroids (TCS) over short periods (4 weeks) in clinically clear appearing skin leads to marked epidermal thinning, altered vasculature, and disrupted collagen structure. A recent review provides a comprehensive appraisal of clinical data relating to several inflammatory skin conditions and the skin atrophy induced from long-term treatment with TCS. The report suggests a relationship between the dose, frequency, duration and anatomical area of application of TCS with the degree of atrophy, and proposes that clinically relevant skin atrophy is more likely to occur from chronic long-term (including intermittent) use of TCS rather than short-term reactive use. Subclinical changes may mark the progression toward clinical adverse effects of TCS misuse, including for example, striae and telangiectasia. Further characterisation of these clinically significant skin changes by OCT is required to inform the understanding of the scale of changes in skin microstructure required to yield clinically significant effects. To do this, researchers also need a robust understanding of healthy skin microstructure.

There are a number of adverse effects associated with TCS use, where used inappropriately or excessively. These adverse effects include hypopigmentation, hypertrichosis, telangiectasia, infection, perioral dermatitis, and atrophy. Usually, these adverse effects are thought to be reversible, but excessive skin atrophy can induce striae atrophicae, which is irreversible. Rarely, systemic absorption can occur due to excessive or long-term use of high-potency TCS, affecting the hypothalamic-pituitary adrenal axis response. However, the risks of TCS-induced Adverse events (AE) can be minimised by using the right dose for limited periods of time (measured in weeks). Epidermal thickness appears to return to normal values within a few weeks after stopping TCS treatment. Parents and carers of AD patients can develop steroid phobia from TCS adverse effects due misinformation from the internet, social media and mixed messages delivered by medical professionals such as GPs, pharmacists or dermatologists who have left clinical practice. This places a significant burden on healthcare workers and caregivers due to underutilisation of TCS, resulting in uncontrolled AD with multiple flare-ups that may require systemic treatment. Further research into the conditions of TCS AEs is required to clarify confusion about their use and enable healthcare professionals (HCPs) to both optimise their safe use and alay patient fears. It is important to educate and train the patient on how to apply the right amount of TCS with the right frequency for each part of the body. Because TCS vary in potency, their safety profiles vary too. According to the British National Formulary (BNF) all topical corticosteroids share side-effects of which some are common or very common (skin reactions, telangiectasia), rare or very rare (adrenal suppression, hypertension, skin depigmentation; may be reversible), and some have unknown frequencies (local reaction, vasodilation). In addition to the major side-effects common to all TCS there are more specific ones for each class and product.

Psychological stress has been shown to exert negative effects on the skin including impaired skin barrier function, loss of stratum corneum integrity and altered immunity. These effects are mediated through the stress-induced hormone cortisol (an endogenously produced steroid). This suggests that a person's stress level and associated cortisol level may be a factor in determining their resting epidermal structure. In fact, the atrophic effects of topically applied corticosteroids (synthetic cortisol derivatives) on the skin demonstrates clearly the impact of glucocorticoid receptor activation on epidermal structure. Moreover, stress, resulting in elevated cortisol levels and Hypothalamic-Pituitary-Adrenal (HPA) -axis overactivation is a recognised trigger for atopic dermatitis and contributes to its progression. Given that, the investigators seek to both understand variations in healthy skin structure and the effects of long-term corticosteroid use, understanding the contribution of stress and the body's cortisol level are important factors. Here the investigators will measure cortisol awakening response from saliva and assess participants stress levels using validated scales.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 6 months old.
* Volunteers understand the purpose, modalities, and potential risks of the study.
* Volunteers are able to read and understand English.
* Volunteers are willing to sign the informed consent.
* [Patient cohort only] Patients diagnosed with AD and

  * A recent history of persistent signs (last flare ≥3 months)
  * Currently controlled signs (ISGA 0-1; clear-almost clear)
  * At least 3 months of TCS use (continuous or intermittent, over the last 6 months)

Exclusion Criteria:

* Participants with any of the following on the measurement skin site (acne, suntan, birthmarks, multiple nevi, tattoos, blemishes, or dense body hair that obstruct the test areas).
* Visible signs of eczema/inflammation at the general measurement sites. Excluding sites of specific interest (SSI) which are imaged in addition to the general measurement sites.
* Participants with a condition that in the opinion of the investigator contradicts participation in the study.

[Healthy cohort only] Participants with a history of chronic skin conditions (except acne).

* Participants who have used any medication that could interfere with the trial aim prior to the start of the study (baseline/visit 1).

[Healthy cohort only] Use of TCS at any point during the 6 months before the clinical visit (except hydrocortisone use for ≤4 weeks outside the target areas of skin).

* Use of any topical product on the measurement areas within 24 hours prior to the measurement visit (>6 hours for patients with severe symptoms).
* Volunteers currently participating in an interventional clinical trial.
* Volunteers incapable of giving fully informed consent.
* Volunteers judged by the PI to be inappropriate for the study.

Min Age: 6 Months | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of 150 healthy skin participants will be identified through advertising to the public (local magazines, email lists, and social media). Healthy skin participants will be subdivided into five age groups (≤30 per group):
  1. Children aged 6 months-10 years old.
  2. Adolescents aged 11-24 years.
  3. Adults aged 25-39 years.
  4. Middle age 40-64 years old.
  5. Adults of older age 65+. A separate patient cohort of ≤30 participants will also be recruited via clinic appointments at the Royal Hallamshire Hospital and Sheffield Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
To quantify epidermal thickness in people with healthy skin | Baseline
  To quantify epidermal thickness (µm) at various body locations in people with healthy skin
To determine tissue attenuation coefficient of whole skin | Baseline
  To determine tissue attenuation coefficient (mm-1)of whole skin, including the epidermis and dermis, at various body locations in people with healthy skin
To determine the vascular plexus depth in people with healthy skin | Baseline
  To determine the vascular plexus depth (µm) at various body locations in people with healthy skin
To determine the vascular density/diameter in people with healthy skin | Baseline
  To determine the vascular density/diameter (segments mm2/µm) at various body locations in people with healthy skin
To determine the collagen matrix index in people with healthy skin | Baseline
  To determine the collagen matrix index (AU) at various body locations in people with healthy skin
To determine skin surface roughness in people with healthy skin | Baseline
  To determine skin surface roughness (µm) at various body locations in people with healthy skin

SECONDARY OUTCOMES:
To determine the effect of sex on epidermal thickness in people with healthy skin | Baseline
  To determine the effect of sex on epidermal thickness (µm) at various body locations in people with healthy skin
To determine the effect of sex on tissue attenuation coefficient in people with healthy skin | Baseline
  To determine the effect of sex on tissue attenuation coefficient (mm-1) at various body locations in people with healthy skin
To determine the effect of sex on vascular plexus depth in people with healthy skin | Baseline
  To determine the effect of sex on vascular plexus depth (µm) at various body locations in people with healthy skin
To determine the effect of sex on vascular density/diameter in people with healthy skin | Baseline
  To determine the effect of sex on vascular density/diameter (segments mm2/µm) at various body locations in people with healthy skin
To determine the effect of sex on collagen matrix index in people with healthy skin | Baseline
  To determine the effect of sex on collagen matrix index (AU) at various body locations in people with healthy skin
To determine the effect of sex on skin surface roughness in people with healthy skin | Baseline
  To determine the effect of sex on skin surface roughness (µm) at various body locations in people with healthy skin
To determine the effect of ethnicity on epidermal thickness in people with healthy skin | Baseline
  To determine the effect of ethnicity on epidermal thickness (µm) at various body locations in people with healthy skin
To determine the effect of ethnicity on tissue attenuation coefficient in people with healthy skin | Baseline
  To determine the effect of ethnicity on tissue attenuation coefficient (mm-1) at various body locations in people with healthy skin
To determine the effect of ethnicity on vascular plexus depth in people with healthy skin | Baseline
  To determine the effect of ethnicity on vascular plexus depth (µm) at various body locations in people with healthy skin
To determine the effect of ethnicity on vascular density/diameter in people with healthy skin | Baseline
  To determine the effect of ethnicity on vascular density/diameter (segments mm-1/µm) at various body locations in people with healthy skin
To determine the effect of ethnicity on collagen matrix index in people with healthy skin | Baseline
  To determine the effect of ethnicity on collagen matrix index (AU) at various body locations in people with healthy skin
To determine the effect of ethnicity on skin surface roughness in people with healthy skin | Baseline
  To determine the effect of ethnicity on skin surface roughness (µm) at various body locations in people with healthy skin
To determine the relationship between skin structure and function in healthy skin | Baseline
  To determine the relationship between skin structure and function in healthy skin (association between structural metrics and transepidermal water loss (TEWL).
To determine the relationship between skin structure and stress | Baseline
  To determine the relationship between skin structure and stress (assessed as perceived stress and salivary cortisol levels).
To quantify epidermal thickness in patients with atopic dermatitis | Baseline
  To quantify epidermal thickness (µm) at various body locations in patients with atopic dermatitis
To determine tissue attenuation coefficient in patients with atopic dermatitis | Baseline
  To determine tissue attenuation coefficient (mm-1) at various body locations in patients with atopic dermatitis
To determine vascular plexus depth in patients with atopic dermatitis | Baseline
  To determine vascular plexus depth (µm) at various body locations in patients with atopic dermatitis
To determine vascular density/diameter in patients with atopic dermatitis | Baseline
  To determine vascular density/diameter (segments mm-1/µm) at various body locations in patients with atopic dermatitis
To determine collagen matrix index in patients with atopic dermatitis | Baseline
  To determine collagen matrix index (AU) at various body locations in patients with atopic dermatitis
To determine skin surface roughness in patients with atopic dermatitis | Baseline
  To determine skin surface roughness (µm) at various body locations in patients with atopic dermatitis

OTHER OUTCOMES:
To discuss the feasibility of conducting a larger study to ascertain the real-world impact of long-term TCS use. | Baseline
  To discuss the feasibility of conducting a larger study to ascertain the real-world impact of long-term TCS use. This is not a quantitative outcome, rather a discussion of practicalities.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Cork, Professor, Principal Investigator — University of Sheffield
Locations (1):
- Royal Hallamshire Hospital, Sheffield Teaching Hospitals NHS FT, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No